CLINICAL TRIAL: NCT00100841
Title: Phase II Trial of FOLFOX6, Bevacizumab and Cetuximab in Patients With Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03006; NCI-6490 (Other: CTEP ID); N01CM62201 (NIH); N01CM62204 (NIH)
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2013-07

CONDITIONS: Adenocarcinoma of the Rectum; Mucinous Adenocarcinoma of the Colon; Recurrent Colon Cancer; Recurrent Rectal Cancer; Signet Ring Adenocarcinoma of the Colon; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms | interventions — Cetuximab; Bevacizumab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): Patients receive cetuximab IV over 60-120 minutes on day 1 in weeks 1-8. Patients also receive bevacizumab IV over 30-90 minutes, oxaliplatin IV over 2 hours, and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 48 hours on days 1 and 2 of weeks 1, 3, 5, and 7. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cetuximab; Biological: bevacizumab; Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil

INTERVENTIONS:
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU

SUMMARY:
Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab and cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of colorectal cancer by blocking blood flow to the tumor. Giving combination chemotherapy together with bevacizumab and cetuximab may kill more tumor cells. This phase II trial is studying how well giving combination chemotherapy together with bevacizumab and cetuximab works in treating patients with stage IV colorectal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, feasibility of administration, response rates and progression free survival among chemotherapy naïve patients with advanced colorectal cancer treated with FOLFOX6 plus bevacizumab and cetuximab (FBC).

II. To determine the survival of patients with advanced colorectal cancer treated with FBC.

III. To determine the safety of the current regimen in selected patients who have had prior MoAb therapy.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV over 60-120 minutes on day 1 in weeks 1-8. Patients also receive bevacizumab IV over 30-90 minutes, oxaliplatin IV over 2 hours, and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 48 hours on days 1 and 2 of weeks 1, 3, 5, and 7. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 40-67 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum which is beyond the scope of surgical resection (MEDRA code:"Colorectal neoplasms malignant","Colorectal cancer stage IV","10010035")
* Measurable disease,
* Life expectancy of greater than 3 months
* ECOG performance status =< 1
* Leukocytes >= 3,500/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 150,000/uL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits
* Patients may not have received prior therapy with bevacizumab or cetuximab
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to radiotherapy administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to any of the agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating women
* Serious or non-healing wound, ulcer or bone fracture
* Invasive procedures defined as follows:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 therapy
  * Anticipation of need for major surgical procedures during the course of the study
  * Core biopsy within 7 days prior to D1 therapy
* If a patient is on full-dose anticoagulants, the following criteria should be met for enrollment:

  * The subject must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin or on stable dose of LMW heparin
  * The subject must not have active bleeding or pathological conditions that carry high risk of bleeding (e.g. tumor involving major vessels, known varices)
* Active infection requiring parental antibiotics on D1
* Proteinuria at baseline; subjects unexpectedly discovered to have >= 1+ proteinuria will undergo a 24-hour urine collection, which will be < 1000 mg protein/ 24 hours to be allowed participation in the study
* No currently active second malignancy other than non-melanoma skin cancer or carcinoma in-situ of the cervix; patients are not considered to have a "currently active" malignancy if they have completed therapy and have no evidence of recurrence for at least 5 years
* Patients with clinically significant cardiovascular disease:

  * Uncontrolled hypertension
  * Myocardial infarction or unstable angina < 6 months prior to registration
  * New York heart association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, unstable angina pectoris
  * Grade II or greater peripheral vascular disease
  * CVA within 6 months of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2004-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allyson Ocean, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Result] Ocean AJ, Polite B, Christos P, Horvath L, Hamilton A, Matulich D, Chen HX, Sparano JA, Kindler HL. Cetuximab is associated with excessive toxicity when combined with bevacizumab Plus mFOLFOX6 in metastatic colorectal carcinoma. Clin Colorectal Cancer. 2010 Dec;9(5):290-6. doi: 10.3816/CCC.2010.n.042. PMID 21208843

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 67 patients were enrolled from between December 2004 and November 2006
Pre-assignment Details: One patient was enrolled but never started treatment
Period: Overall Study
Arm/Group | Treatment (Combination Chemotherapy)
Started | 66
Completed | 66
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 66
Age, Continuous [Median (Full Range); unit: years] | 57 [27 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 35
Race/Ethnicity, Customized [Number; unit: participants]
  White | 51
  Black | 10
  Asian | 2
  Hispanic | 3

OUTCOME MEASURES:

1. Primary Outcome: Severe Adverse Event (SAE) Rate
Description: The primary objective is to evaluate safety in all treated patients specifically the rate of serious adverse events which were defined as grade 5 events, grade 4 hemorrhage or thrombosis or bowel perforation
Time Frame: The duration of the study
Population: 66 patients treated with cetuximab
Measure: Number; unit: participants
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 66
participants
  Grade 5 Death | 2
  Grade 4 venous thrombosis | 2

2. Primary Outcome: Progression Free Survival Rate
Time Frame: From randomization to the first documented disease progression
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 38
months | 9.6 [9.5 to 12.2]

ADVERSE EVENTS:
Arm/Group | Treatment (Combination Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 54/66
Other Adverse Events (participants affected / at risk) | 63/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Combination Chemotherapy) (N=66)
Hemoglobin (anemia) (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 15 (15)
Catheter-related infection (Infections and infestations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Ungual (nails) infection (Infections and infestations) | 1 (1)
Cardiopulmonary-restrictive (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Fatigue (General disorders) | 9 (9)
Cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 2 (2)
Alanine transaminase (Investigations) | 2 (2)
Aspartate transaminase (Investigations) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Oral mucositis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 3 (3)
Neuropathy: Sensory (Nervous system disorders) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Combination Chemotherapy) (N=66)
Eye infection (Infections and infestations) | 6 (6)
Upper airway infection (Infections and infestations) | 5 (5)
Upper tract infection (Infections and infestations) | 3 (3)
Hypertension (Vascular disorders) | 10 (10)
Hemorrhage: nose (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Hemorrhage: lower gastrointestinal (Gastrointestinal disorders) | 7 (7)
Hemorrhage: urine (Renal and urinary disorders) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (11)
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 16 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less